CLINICAL TRIAL: NCT01697800
Title: A Phase II Trial of Tadalafil in Patients With Squamous Cell Carcinoma of the Upper Aero Digestive Tract
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: J1247; 2P50DE019032 (NIH); NA_00073880 (Other: JHMIRB)
Record Dates: First submitted 2012-09-28; First posted 2012-10-02 (Estimated); Results first posted 2020-02-28 (Actual); Last update posted 2020-02-28 (Actual); Status verified 2020-02

CONDITIONS: Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Tadalafil

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Patients received placebo capsules for 2 weeks prior to standard of care treatment and continued for 3 months post standard of care treatment
  Interventions: Drug: Placebo
- Tadalafil (Active Comparator): Patients received 20 mg tadalafil capsules for 2 weeks prior to standard of care treatment and continued for 3 months post standard of care treatment
  Interventions: Drug: Tadalafil

INTERVENTIONS:
Drug: Tadalafil
  Other Names: Cialis
  Arms: Tadalafil
Drug: Placebo
  Arms: Placebo

SUMMARY:
Head and neck squamous cell carcinoma (HNSCC) is a lethal solid malignancy with 5 year survival estimates of approximately 50%, and is associated with a high rate of systemic immune impairment as well as evasion of a tumor specific immune response. Preclinical and clinical data have shown that phosphodiesterase 5 (PDE5) inhibitors (tadalafil) can be used to augment immune function in HNSCC patients through inhibition of the cancer-induced myeloid derived suppressor cells (MDSCs).

A multi site phase II, randomized, prospective, biomarker endpoint trial to determine optimum timing and design of PDE5 antitumor immunotherapy (tadalafil) in conjunction with conventional therapy for HNSCC.

40 patients with biopsy proven HNSCC will be randomized to receive tadalafil (n=25) or placebo (n=15) for at least 10-14 days before starting conventional therapy and continuing until 90 days after completion of conventional therapy. Tumor-specific T cell responses will be assessed using HNSCC cell lines, in blood collected before initiation of tadalafil/placebo and at 60 and 90 days after completion of conventional therapy. Number and function of MDSC and Treg cells will be assessed before and at 60 and 90 days after completion of conventional therapy. Prevnar 13® vaccine will be administered 10-14 days after commencing tadalafil/placebo (before conventional therapy begins) and again at 60 days after completion of conventional therapy. Vaccine-specific responses assessed at 60 and 90 days post-conventional therapy will be used to measure the ability of tadalafil to augment immune response to vaccine.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥21 years
2. Histologically confirmed, previously untreated invasive head and neck squamous cell carcinoma OR histologically confirmed not yet treated recurrent head and neck squamous cell carcinoma (must be at least 3 months after diagnosis and completion of treatment for primary disease or last recurrence). Patients may have local Stage I or II, or locoregionally advanced HNSCC Stage III or IV of the oral cavity, oropharynx, larynx, hypopharynx, or unknown primary, but no metastatic disease; Intent to treat with primary radiotherapy +/-chemotherapy
3. Disease location amenable to biopsy in outpatient clinical setting or operative biopsy within routine accepted schedule and practice of clinical care
4. Eastern Cooperative Oncology Group (ECOG) performance status 0-1
5. Required laboratory data (to be obtained within 2 weeks of initiation):

   * Platelets > 75,000/mm³
   * Calculated Creatinine Clearance (CRCL)> 60 mL/min
   * Total serum bilirubin < 1.5 mg/dL
6. Willingness and ability to give signed written informed consent.

Exclusion Criteria:

1. Medical contraindication to biopsy of target lesion
2. Intercurrent illness likely to prevent protocol therapy or conventional planned therapy
3. Prior daily use of tadalafil or other long-acting PDE5 inhibitors for one month or greater
4. Known severe hypersensitivity to tadalafil or any of the excipients of this product
5. Current treatment with nitrates
6. Current systemic treatment with a potent cytochrome P450 3A4 (CYP3A4) inhibitor such as ketoconazole or ritonavir
7. History of hypotension and/or blindness during prior treatment with tadalafil or other PDE5 inhibitors
8. Prior history of non-arterial ischemic optic retinopathy
9. Prior adverse reaction to diphtheria vaccine
10. Pregnant or breastfeeding; a negative pregnancy test is required within 14 days of randomization for all women of childbearing potential.
11. Concurrent malignancy or a history of previous malignancy treated with curative therapy within the last 3 months (other than squamous/basal cell cancer of the skin or cervical cancer), for which the survival prognosis is < 5 years
12. Treatment with a non-approved or investigational drug within 30 days before visit 1
13. Incomplete healing from previous oncologic or other major surgery
14. As judged by the investigator, any evidence of severe or uncontrolled systemic disease (e.g., unstable or uncompensated respiratory, cardiac, hepatic, or renal disease)
15. Evidence of any other significant clinical disorder or laboratory finding that makes it undesirable for the subject to participate in the trial
16. History of significant hypotensive episode requiring hospitalization
17. History of acute myocardial infarction within prior 3 months, uncontrolled angina, uncontrolled arrhythmia, or uncontrolled congestive heart failure
18. History of any of the following cardiac conditions:

    I. Angina requiring treatment with long-acting nitrates II. Angina requiring treatment with short-acting nitrates within 90 days of planned tadalafil administration III. Unstable angina within 90 days of visit 1 (Braunwald 1989) IV. Positive cardiac stress test without documented evidence of subsequent, effective cardiac intervention
19. History of any of the following coronary conditions within 90 days of planned tadalafil administration:

    I. Myocardial Infarction II. Coronary artery bypass graft surgery III. Percutaneous coronary intervention (for example, angioplasty or stent placement) IV. Any evidence of heart disease (NYHA≥Class III as defined in Protocol Attachment LVHG.3) within 6 months of planned tadalafil administration
20. Prior chronic immune suppressive state (AIDS, immunosuppressive therapy)

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-09; Primary Completion 2014-07-14 (Actual); Study Completion 2014-07-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zubair Khan, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Guo T, Califano JA. Molecular biology and immunology of head and neck cancer. Surg Oncol Clin N Am. 2015 Jul;24(3):397-407. doi: 10.1016/j.soc.2015.03.002. Epub 2015 Apr 20. PMID 25979390

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Tadalafil
Started | 15 | 25
Completed | 15 | 24
Not Completed | 0 | 1
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Tadalafil | Total
Number analyzed (Participants) | 15 | 25 | 40
Age, Customized [Count of Participants; unit: Participants]
  18-99 years | 15 | 25 | 40
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 14 | 23 | 37
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 4 | 6
  White | 13 | 21 | 34
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15 | 25 | 40

OUTCOME MEASURES:

1. Primary Outcome: Change in Immune Response After Tadalafil Administration
Time Frame: Baseline and 120-150 Days
Population: Blood samples were collected. However, the samples were not analyzed and hence no data were generated.
Arm/Group | Placebo | Tadalafil
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Placebo | Tadalafil
All-Cause Mortality (participants affected / at risk) | 0/15 | 1/25
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/25
Other Adverse Events (participants affected / at risk) | 0/15 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No